CLINICAL TRIAL: NCT07088432
Title: Intravenous Dexamethasone for Prolonging the Sensory Block Duration of Spinal Anesthesia: A Randomized Controlled Trial
Brief Title: Intravenous Dexamethasone for Prolonging Sensory Block in Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Kamel ben Fadhel, Professor, Department of Anesthesiology and Intensive Care, Habib Thameur Hospital, Tunis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HTHEC-2023-26
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Spinal Anesthesia; Postoperative Pain Management; Dexamethasone; Pelvic Surgery; Urologic Surgery; Proctologic Surgery
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, randomized controlled trial with 1:1 allocation
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient, anesthesia provider, surgeon, and outcome assessor were all blinded to group allocation. The syringes were prepared by a resident not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Dexamethasone Group (Experimental): Participants in this arm received 8 mg of intravenous dexamethasone (2 mL) 5 minutes before spinal anesthesia. The spinal anesthesia was performed with 12.5 mg of 0.5% hyperbaric bupivacaine combined with 2.5 µg of sufentanil. The purpose was to evaluate whether intravenous dexamethasone prolongs the duration of sensory and motor block and improves postoperative analgesia.
  Interventions: Drug: Dexamethasone
- Placebo Group (Placebo Comparator): Participants in this arm received 2 mL of isotonic saline intravenously 5 minutes before spinal anesthesia. The spinal anesthesia was performed identically to the intervention group (12.5 mg of hyperbaric bupivacaine + 2.5 µg sufentanil). This arm served as the control group for evaluating the effects of dexamethasone.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Single intravenous injection of 8 mg dexamethasone (2 mL) administered 5 minutes before spinal anesthesia. This intervention was tested for its effect on prolonging the duration of sensory and motor blocks induced by hyperbaric bupivacaine combined with sufentanil. The drug was administered under sterile conditions by an anesthesiologist blinded to group allocation.
  Arms: Intravenous Dexamethasone Group
Drug: Placebo — Single intravenous injection of 2 mL isotonic saline (0.9% NaCl) administered 5 minutes before spinal anesthesia. This placebo was used to mimic the dexamethasone injection in the control group. The preparation, volume, and timing were identical to the intervention group to maintain blinding. The saline was administered under sterile conditions by an anesthesiologist blinded to group allocation.
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to learn if intravenous dexamethasone can help prolong the effect of spinal anesthesia in adults having elective pelvic, urologic, or proctologic surgery. The study also looks at whether dexamethasone improves pain control after surgery and whether it causes any side effects.

The main questions it aims to answer are:

Does intravenous dexamethasone increase how long the spinal anesthesia lasts?

Does it reduce the need for pain medications after surgery?

Does it cause more or fewer side effects compared to a placebo?

In this study:

Participants were randomly assigned to receive either 8 mg of intravenous dexamethasone or a placebo (salt water).

All participants received standard spinal anesthesia with bupivacaine and sufentanil.

Researchers measured how long the spinal anesthesia lasted and when the first pain medication was needed after surgery.

Participants were monitored for side effects such as low blood pressure, nausea, vomiting, and slow heart rate.

Surgeon satisfaction with anesthesia quality was also recorded.

Participants did not receive any additional procedures beyond routine care. The study found that dexamethasone helped prolong the spinal anesthesia and delayed the need for pain relief, without increasing side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 80 years

ASA physical status I or II

Scheduled for elective pelvic surgery under spinal anesthesia (urologic, inguinal, or proctologic procedures)

Provided informed consent

Exclusion Criteria:

* Known allergy to dexamethasone or local anaesthetics

Contraindications to spinal anesthesia

Neurological diseases

Chronic use of corticosteroids or immunosuppressants

BMI > 40 kg/m²

Refusal to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block | From the time of spinal injection until sensory regression to L1 dermatome (up to 4 hours postoperatively)
  The duration of the sensory block was defined as the time from intrathecal injection of the local anesthetic until regression of sensory level to the L1 dermatome, as assessed by pinprick test every 15 minutes postoperatively. This endpoint was selected to evaluate the effect of intravenous dexamethasone on prolonging the duration of spinal anesthesia.

SECONDARY OUTCOMES:
Duration of motor block | From the time of spinal injection until modified Bromage score = 3 (up to 4 hours postoperatively)
  The duration of the motor block was defined as the time from intrathecal injection until achieving a modified Bromage score of 3, which corresponds to partial motor recovery (able to move knees). The modified Bromage score was assessed every 15 minutes postoperatively. This measure was used to assess whether intravenous dexamethasone prolongs motor block following spinal anesthesia.
Time to first analgesic request | From spinal injection until VAS score ≥ 3 and first analgesic request (up to 6 hours postoperatively)
  Time from intrathecal injection to the first request for postoperative analgesia, defined as the moment when the patient reported a pain score ≥ 3 on a visual analog scale (VAS, 0-10). This was recorded in minutes starting from the time of spinal anesthesia. The aim was to assess whether intravenous dexamethasone prolongs the duration of effective postoperative analgesia.
Incidence of adverse events | From spinal injection until the end of surgery
  Adverse events occurring during the surgical procedure were systematically recorded. These included hypotension (systolic BP < 90 mmHg), bradycardia (HR < 50 bpm), nausea, vomiting, pruritus, and any signs of discomfort or neurological complications. All events were recorded as present or absent and compared between the dexamethasone and placebo groups to assess the safety profile of intravenous dexamethasone during spinal anesthesia.
Surgeon satisfaction score | Immediately after the end of surgery
  Surgeon satisfaction with the quality of intraoperative anesthesia was assessed using a binary score (Satisfied / Not satisfied). The evaluation was based on intraoperative conditions such as patient immobility, comfort, and adequacy of anesthesia. The rating was collected at the end of surgery to compare the perceived quality between the dexamethasone and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Samia Arfaoui, Medical Doctor, Study Director — Habib Thameur Hospital; Kamel Ben Fadhel, Medical Doctor, Study Chair — Habib Thameur Hospital
Locations (1):
- Habib Thameur Hospital, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided